CLINICAL TRIAL: NCT00476307
Title: A Phase III Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix™ (Influsplit SSW®) 2007/2008 in People Aged 18 Years or Above
Brief Title: Immunogenicity and Reactogenicity of Fluarix™ (Influsplit SSW®) 2007/2008 in People 18 Years Old or Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110221
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Flu vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Fluarix™/Influsplit SSW® 2007/2008

SUMMARY:
This study is designed to test the immunogenicity and reactogenicity of the Fluarix™/Influsplit SSW® containing the influenza strains recommended for the 2007-2008 season.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 years or above;
* Non-childbearing or using adequate contraception;
* Written informed consent obtained from the subject.

Exclusion Criteria:

Subjects must not:

* Participate in a trial or using non-registered product;
* Use immunosuppressants, blood products, or another influenza vaccine during study;
* Have virologically confirmed influenza within 1 year;
* Have allergic or acute disease;
* Have unstabilized serious chronic disease;
* Be a lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Immune response 21 days post vaccination

SECONDARY OUTCOMES:
Safety: solicited local and general symptoms, unsolicited symptoms, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110221 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register